CLINICAL TRIAL: NCT06660134
Title: Strict Weight Management and Glycemic Control Based on Glucagon-like Peptide-1 (GLP-1) Receptor Agonist Treatment VS. Conventional Antidiabetic Drugs for Ablation Outcomes in Overweight or Obese Patients with Type 2 Diabetes and Atrial Fibrillation
Brief Title: Strict Weight Management Based on GLP-1 RA for Ablation Outcomes in Overweight or Obese Patients with T2DM and AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: The Third Affiliated Hospital of Anhui Medical University (Unknown); The Second People's Hospital of Anhui Province (Other); Hefei Second People's Hospital (Unknown)
Responsible Party: Principal Investigator, Xu Liu, Dr, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWGLP-AF
Record Dates: First submitted 2024-09-27; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Atrial Fibrillation (AF)
Keywords: Catheter ablation; Glucagon-like Peptide-1 receptor agonist; Atrial fibrillation; overweight; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atrial Fibrillation; Overweight; Obesity | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strict Weight Reduction Intervention Group (Experimental): In addition to the routine use of Antiarrhythmic Drugs (AADs) and anticoagulants, the strict weight reduction intervention group also uses GLP-1 receptor agonists for glycemic control and weight loss according to guidelines. This group receives a structured weight loss program, regular nutritional advice in accordance with current guidelines, and physical training assistance over a 12 month period. The intervention plan aims for a total weight loss of 10 kilograms while using GLP-1 receptor agonists.
  Interventions: Drug: Glucagon-like peptide-1 receptor agonists (GLP 1 RA)
- Standard Care Group (Active Comparator): Receives standard glycemic control treatment for diabetes and follows the recommended anticoagulant and antiarrhythmic drug regimens post ablation.
  Interventions: Drug: Glucagon-like peptide-1 receptor agonists (GLP 1 RA)

INTERVENTIONS:
Drug: Glucagon-like peptide-1 receptor agonists (GLP 1 RA) — In addition to the routine use of Antiarrhythmic Drugs (AADs) and anticoagulants, the strict weight reduction intervention group also uses GLP-1 receptor agonists for glycemic control and weight loss according to guidelines. This group receives a structured weight loss program, regular nutritional advice in accordance with current guidelines, and physical training assistance over a 12-month period. The intervention plan aims for a total weight loss of 10 kilograms while using GLP-1 receptor agonists.

SUMMARY:
Objective To compare, in patients with Type 2 Diabetes Mellitus (T2DM) and Atrial Fibrillation (AF) undergoing radiofrequency ablation (RFA), whether strict weight management and glycemic control based on Glucagon-like Peptide-1 (GLP-1) receptor agonist treatment reduces the recurrence rate of atrial arrhythmias and rehospitalization rates for cardiac diseases compared to conventional post-procedural management (antiarrhythmic drugs and anticoagulants) and general antidiabetic drugs (excluding GLP-1 receptor agonists).

Study Design

This trial randomly divides participants into two groups:

The GLP-1 receptor agonist treatment-based strict weight management and glycemic control group.

The conventional treatment group

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years. Symptomatic atrial fibrillation (AF) that has been ineffective or intolerable to at least one Class I or III antiarrhythmic drug.

Diagnosed with Type 2 Diabetes Mellitus. Body Mass Index (BMI) greater than 25 kg/m². Ability to understand the purpose of the trial, willingness to participate, and signing of the informed consent form.

Exclusion Criteria:

Permanent atrial fibrillation (failed cardioversion or episode duration >12 months).

Previous history of AF ablation treatment. History of acute coronary syndrome or percutaneous coronary intervention within 6 months prior to enrollment.

History of implantation of an implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy (CRT).

History of stroke or transient ischemic attack within 6 months prior to enrollment.

Severe organic heart disease, including moderate to severe mitral regurgitation or stenosis, previous myocardial infarction, hypertrophic cardiomyopathy, etc.

History of left atrial appendage occlusion or planned for one-stop AF ablation and left atrial appendage occlusion.

Pregnant, breastfeeding, or planning to become pregnant. Significant bleeding tendency precluding post-procedural systemic anticoagulation.

Contraindications to oral hypoglycemic agents such as SGLT2 inhibitors or GLP-1 receptor agonists.

Presence of left atrial thrombus identified before the procedure. Previous cardiac surgery (valve repair/replacement, coronary artery bypass grafting).

Unable to perform physical exercise due to illness or disability. Significant hyperthyroidism or hypothyroidism. Drug abuse or chronic alcoholism. Comorbidity with other serious illnesses with an expected survival less than 12 months.

Any condition that does not align with the best interest of the subject. Other conditions determined by the investigator as unsuitable for inclusion in this study, such as psychiatric disorders or psychological impairments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation (AF), atrial flutter (AFL), or atrial tachycardia events lasting ≥30 seconds occurring from the end of a 3-month blanking period post-procedure up to 12 months of follow-up. | at least 12 months of follow-up, beyond the initial 3-month blanking period

SECONDARY OUTCOMES:
Changes in Body Mass Index (BMI) from baseline to 12 months. | at least 12 months of follow-up, beyond the initial 3 month blanking period
  Combine weight and height, and report the Body Mass Index (BMI) in units of kilograms per square meter (kg/m²).
Quality of life assessments. | at least 12 months of follow-up, beyond the initial 3-month blanking period
  The quality of life and cardiac function of the subjects were assessed using the World Health Organization Quality of Life (WHOQOL-100) questionnaire.
Complications associated with AF ablation and serious adverse events (such as rehospitalizations, cardiovascular rehospitalizations) occurring during the study period. | at least 12 months of follow-up, beyond the initial 3-month blanking period
Quality of life assessments | at least 12 months of follow-up, beyond the initial 3-month blanking period
  Quality of life assessments were conducted within at least 12 months of follow-up using measures such as the AF6.
Quality of life assessments | at least 12 months of follow-up, beyond the initial 3-month blanking period
  Quality of life assessments were conducted using the AFEQT (Atrial Fibrillation Effect on Quality of Life) questionnaire.
Psychological distress | at least 12 months of follow-up, beyond the initial 3-month blanking period
  Psychological distress was assessed using the HADS (Hospital Anxiety and Depression Scale).
Functional status | at least 12 months of follow-up, beyond the initial 3 month blanking period
  Functional status was assessed using the CCS-SAF (Canadian Cardiovascular Society - Self-Assessed Functioning scale).
quality of life | at least 12 months of follow-up, beyond the initial 3-month blanking period
  The quality of life and cardiac function of the subjects were assessed using the New York Heart Association (NYHA) functional classification.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Liu, Dr, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided